CLINICAL TRIAL: NCT00000957
Title: A Phase I Multicenter Clinical Trial to Evaluate the Safety and Immunogenicity of Vaccinia Derived HIV-1 Recombinant Envelope Glycoprotein (gp160) of Human Immunodeficiency Virus: Evaluation of Accelerated Schedules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immuno-US (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 004B; 10545 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV-1; Drug Evaluation; HIV Envelope Protein gp160; Drug Administration Schedule; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)

SUMMARY:
To evaluate the safety and immune response to vaccinia-derived HIV-1 recombinant envelope glycoprotein (gp160) using an accelerated dosage schedule; to evaluate duration of antibody response and its relationship to the dose and frequency of inoculation.

Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure for AIDS. It is likely that ultimate control of the disease depends on the development of safe and effective vaccines against HIV.

DETAILED DESCRIPTION:
Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure for AIDS. It is likely that ultimate control of the disease depends on the development of safe and effective vaccines against HIV.

Thirty healthy adult volunteers without identifiable high-risk behavior for HIV-1 are randomly assigned to receive vaccination with gp160 (50 mcg) according to one of the following schedules: Group 1 receives vaccine on days 0, 28, 56, and 140 and placebo on days 84 and 112; Group 2 receives vaccine on days 0, 28, 56, 84, and 112 and placebo on day 140. Subjects are followed for 1 year after the last injection. Per 05/13/94 amendment, 10 subjects at the St. Louis University site receive an additional boost 18-24 months after the last injection.

ELIGIBILITY:
Inclusion Criteria

Patients must be:

* Normal, healthy, HIV-negative adults who fully comprehend the purpose and details of the study.
* Available for 1 year of follow-up.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* They or their sexual partners have identifiable high-risk behavior for HIV infection.
* Positive syphilis serology (e.g., VDRL).
* Positive for circulating hepatitis B antigen.

Patients with the following prior conditions are excluded:

* History of positive PPD (tuberculin test).
* History of immunodeficiency or chronic illness.
* Evidence of depression or under treatment for psychiatric problems during the past year.

Prior Medication:

Excluded:

* Immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood transfusions or cryoprecipitates within the past 6 months.

Risk Behavior: Excluded:

* High-risk behavior for HIV infection.
* History of intravenous drug use.
* More than one sexual partner in the last 6 months.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Study Completion 1993-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair
Locations (3):
- United States (3):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - JHU AVEG, Pittsburgh, Pennsylvania
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee

REFERENCES:
- [Background] Keefer MC, Wolff M, Gorse GJ, Graham BS, Corey L, Clements-Mann ML, Verani-Ketter N, Erb S, Smith CM, Belshe RB, Wagner LJ, McElrath MJ, Schwartz DH, Fast P. Safety profile of phase I and II preventive HIV type 1 envelope vaccination: experience of the NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1997 Sep 20;13(14):1163-77. doi: 10.1089/aid.1997.13.1163. PMID 9310283
- [Background] Gorse GJ, Schwartz DH, Graham BS, Matthews TJ, Stablein DM, Frey SE, Belshe RB, Clements ML, Wright PF, Eibl M, et al. HIV-1 recombinant gp160 vaccine given in accelerated dose schedules. NIAID AIDS Vaccine Clinical Trials Network. Clin Exp Immunol. 1994 Nov;98(2):178-84. doi: 10.1111/j.1365-2249.1994.tb06122.x. PMID 7955519
- [Background] Gorse GJ, Patel GB, Newman FK, Mandava M, Belshe RB. Recombinant gp160 vaccination schedule and MHC HLA type as factors influencing cellular responses to HIV-1 envelope glycoprotein. NIAID AIDS Vaccine Clinical Trials Network. Vaccine. 1995 Sep;13(13):1170-9. doi: 10.1016/0264-410x(95)00020-2. PMID 8578800